CLINICAL TRIAL: NCT00698204
Title: Cyclooxygenase-2 Inhibition in Radiation-Induced Oral Mucositis
Brief Title: Cox-2 Inhibition in Radiation-induced Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Pfizer (Industry)
Responsible Party: Principal Investigator, Rajesh Lalla, Associate Professor, Oral Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 03 -157- 2; GCRC 487 (Other: UCHC Clinical Research Center); COXAON-0509-150 (Other: Pfizer, Inc.); K23DE016946-05 (NIH)
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Oral Mucositis
Keywords: Mucositis; Head and Neck Cancer; Head and Neck Neoplasms; Stomatitis
MeSH Terms: conditions — Stomatitis; Mucositis; Head and Neck Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I- Celecoxib (Experimental)
  Interventions: Drug: celecoxib
- II (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celecoxib — Subject was asked to take celecoxib each day that radiation therapy was given.
  Other Names: Celebrex
  Arms: I- Celecoxib
Drug: placebo — Subject was asked to take placebo each day that radiation therapy was given.
  Arms: II

SUMMARY:
Oral mucositis refers to ulcerative lesions of the oral mucosa that occur due to radiation therapy given for treatment of head and neck cancer. These lesions are painful, compromise nutrition and quality of life and may necessitate interruptions in radiation therapy, thus adversely affecting cancer therapy outcomes. This study examined the use of an anti-inflammatory medicine to reduce pain and severity of oral mucositis.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who will be receiving at least 5000 centigray (cGy) radiation therapy to at least 2 of 14 pre-defined areas in the oral cavity.
* Women of childbearing potential must agree to use a medically accepted form of contraception during the course of the study. Women of childbearing potential must have a documented negative pregnancy test within fourteen days of enrollment in the study.
* Patient's willing and able to provide written informed consent for the study.

Key Exclusion Criteria:

* Patients with known hypersensitivity to celecoxib or other COX-2 inhibitors.
* Patients who have experienced asthma, urticaria, or allergic-type reactions after taking salicylates (e.g. aspirin) or Non-steroidal anti-inflammatory drugs (NSAIDs).
* Patients who have demonstrated allergic-type reactions to sulfonamides.
* Patients with a history of gastric, esophageal, pyloric channel or duodenal ulcer disease or gastrointestinal bleeding.
* Patients with a history of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis) or pancreatic disease.
* Patients with severe hepatic impairment.
* Patients with advanced renal disease.
* Patients with a significant bleeding disorder.
* Patients under the age of 18 or over the age of 75.
* Women who are pregnant or nursing.
* Patients with a history of thromboembolic events including myocardial infarction, pulmonary embolism, deep venous thrombosis, transient ischemic attack and ischemic cerebrovascular accident (stroke).
* Patients who have had coronary angioplasty, coronary artery bypass surgery or another cardiac revascularization procedure.
* Patients with a history of a cardiac arrhythmia requiring anti-arrhythmic therapy, angina pectoris or congestive heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-07; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh V Lalla, DDS, Ph.D, CCRP, Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut

REFERENCES:
- [Derived] Lalla RV, Choquette LE, Curley KF, Dowsett RJ, Feinn RS, Hegde UP, Pilbeam CC, Salner AL, Sonis ST, Peterson DE. Randomized double-blind placebo-controlled trial of celecoxib for oral mucositis in patients receiving radiation therapy for head and neck cancer. Oral Oncol. 2014 Nov;50(11):1098-103. doi: 10.1016/j.oraloncology.2014.08.001. Epub 2014 Aug 21. PMID 25151488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period University of Connecticut Health Center: December 2003 through December 2004 and from March 2006 through June 2011.
  Recruitment period Hartford Hospital: March 2010 thorough June 2011.
Pre-assignment Details: Three participants enrolled in the study but were not randomized. Two did not meet blood test eligibility criteria for randomization (liver function test, renal function test failure) and one withdrew shortly after enrolling, prior to randomization.
Groups:
- I- Celecoxib: celecoxib: Subjects were randomized to take celecoxib each day that radiation therapy was given (6-7 week period).
- II- Placebo: placebo: Subject was randomized to take an identical placebo each day that radiation therapy was given (6-7 week period).
Period: Overall Study
Arm/Group | I- Celecoxib | II- Placebo
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis performed for 40 participants. Per-protocol analysis performed for the period in which individual participants were taking study medication (celecoxib or placebo).
Groups:
- I- Celecoxib: celecoxib: Subject was randomized to take celecoxib each day that radiation therapy was given.
- II- Placebo: placebo: Subject was randomized to take placebo each day that radiation therapy was given.
- Total: Total of all reporting groups
Arm/Group | I- Celecoxib | II- Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 53.15 [34 to 71] | 56.00 [36 to 69] | 54.58 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 17 | 15 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Oral Mucosal Injury Score at Cumulative Radiation Dose of 5000 cGy
Description: Oral Mucositis Assessment Scale (OMAS) was used to assess oral mucosal injury during the period of radiation therapy. This validated scale scores ulceration and erythema independently at nine specified sites in the oral cavity. Ulceration is scored from 0-3 based on size of lesion and erythema is scored from 0-2 based on severity of erythema. The sum of scores is then divided by 9.
  The mean OMAS score at a cumulative radiation dose of 5000 cGy (approximately 5 weeks of treatment) was compared between groups.
Time Frame: 5 weeks from start of radiation therapy (5000 cGy)
Population: Subjects participating in the study as they reached a cumulative dose of 5000 cGy were included. One subject in the celecoxib group withdrew prior to reaching 5000 cGy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I- Celecoxib | II- Placebo
Number analyzed (Participants) | 19 | 20
units on a scale | 1.42 (.67) | 1.36 (.88)

2. Secondary Outcome: Evaluation of Pain Severity at 5000 cGy Radiation
Description: Mean worst pain at 5000 cGy on 0-10 scale, 0 = no pain, 10 = worst pain imaginable
Time Frame: 5 weeks from start of radiation therapy (cumulative dose of 5000 cGy)
Population: Only subjects who were still taking the study drug (celecoxib or placebo) when cumulative radiation dose of 5000 cGy was reached are included in this analysis (19 of 20 in each group were analyzed).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I- Celecoxib | II- Placebo
Number analyzed (Participants) | 19 | 19
units on a scale | 4.47 (2.82) | 3.70 (3.20)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of Informed Consent through 30 days after the last study intervention.
Description: All events reported as serious adverse events resulted in hospitalization of the participant during the period of study participation. All adverse events were reviewed by an independent Data and Safety Monitoring Board (DSMB) and were determined to be unrelated to use of celecoxib.
Arm/Group | I- Celecoxib | II- Placebo
Serious Adverse Events (participants affected / at risk) | 6/20 | 5/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I- Celecoxib (N=20) | II- Placebo (N=20)
Electrolyte abnormality (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 3 (3) | 3 (3)
Myocardial infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — This event was reviewed by the DSMB and was determined to be unrelated to use of celecoxib.
Nausea/vomiting (Gastrointestinal disorders) | 3 (8) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — This event was reviewed by the DSMB and was determined to be unrelated to use of celecoxib.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I- Celecoxib (N=20) | II- Placebo (N=20)
pruritus (Immune system disorders) | 1 (1) | 0 (0) — antibiotic drug reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No